CLINICAL TRIAL: NCT04173650
Title: Mesenchymal Stem Cell Extracellular Vesicles for the Treatment of Recessive Dystrophic Epidermolysis Bullosa Wounds
Brief Title: MSC EVs in Dystrophic Epidermolysis Bullosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aegle Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EB IND
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Dystrophic Epidermolysis Bullosa
Keywords: Exosomes; Extracellular Vesicles
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, open label, randomized, multi-center study, with intra-subject paired- wound control, intended to assess the safety and preliminary efficacy of administering EVs derived from allogeneic MSCs to 10-50 cm2 wounds in RDEB subjects with wounds persisting for at least four weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- AGLE 102 (Experimental): Treatment arm
  Interventions: Drug: AGLE-102

INTERVENTIONS:
Drug: AGLE-102 — Extracellular vesicles from bone marrow derived mesenchymal stem cells - up to six topical administrations
  Other Names: AGLE 102; Control

SUMMARY:
INVESTIGATIONAL PRODUCT: AGLE-102 is an allogeneic extracellular vesicle (EV) product derived from normal donor mesenchymal stem cells (MSCs).

INDICATION AND RATIONALE: The aim of the study is to assess the safety and efficacy of AGLE-102 in the treatment of lesions in subjects with Epidermolysis Bullosa (EB).

STUDY DESIGN: This is a phase 1/2A, randomized, multi-center, study to assess the effectiveness and safety of AGLE-102 on lesions in subjects with EB.

DETAILED DESCRIPTION:
STUDY DESIGN: This is a prospective, open label, randomized, multi-center study, with intra-subject paired wound standard of care control, intended to assess the safety and preliminary efficacy of administering EVs derived from allogeneic MSCs to 10-50 cm2 wounds in RDEB subjects with wounds persisting for at least four weeks.

After providing written informed consent (assent with parental written consent for pediatric subjects) and undergoing screening evaluations, eligible subjects have a single set of paired wounds identified that are determined by either subject/caregiver reporting, medical history or other reliable sources to have been present for a minimum of four weeks. One of each pair is randomized to treatment with EVs in conjunction with standard of care. The other wound of each pair receives standard of care alone, without EV treatment. All wounds on study continue to receive standard of care throughout the study. For the EV treated wounds, up to six administrations of EVs occur approximately two weeks apart over a period of 10 weeks. If the treated wound closes prior to six administrations, no additional doses are given unless the wound reopens during the treatment period, in which case the original retreatment schedule resumes but is not extended. Subjects with wound closure identified at one of the treatment visits should return for all subsequent visits to verify wound closure and assess the scar quality of the wound, unless the closure is identified at the final study visit, in which case no additional visits are required.

Wound closure is determined by complete re-epithelialization that is not subject to re-injury during dressing changes or as a result of normal daily activities (e.g., wearing clothing, eating, sleeping). This is confirmed by the investigator at least two weeks after initial closure (unless closure is identified at the final study visit). At the conclusion of the 10-weektreatment period, the wounds are followed every 4 weeks for a period of 12 weeks. At no time during the study does closure status of the control wound influence the EV treatment or visit schedule.

STUDY OBJECTIVES:

Primary Objectives:

Determine the safety of applying multiple administrations of EVs derived from allogeneic MSCs to 10-50 cm2 RDEB wounds that have persisted for at least four weeks

Determine if EVs plus standard of care can promote wound healing in RDEB subjects compared to standard of care alone control

Secondary Objectives: Determine if there is clinical benefit of applying EVs to RDEB wounds

PLANNED SAMPLE SIZE: 8 subjects will be treated on the protocol with AGLE-102.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 6 months or older at screening.
2. Subjects who have a confirmed diagnosis of DEB based on electron microscopy, immunomapping, or genetic testing. Subjects with severe DEB (e.g., RDEB patients with absent Col VII/no anchoring fibrils) and milder forms of DEB (e.g., RDEB patients with reduced Col VII and/or anchoring fibril levels) are eligible.
3. Presence for at least four weeks of two 10 - 50 cm2 wounds (unroofed EB erosions) at least 4 inches apart that can be considered similar enough in size, wound location and expected healing characteristics to be a matched pair. Neither index wound may have been treated with any local (topical, subcutaneous, etc) or systemic therapeutic other than standard of care treatments described in this protocol (i.e. local or systemic antimicrobials to control infection, topical anesthetic and oral analgesics if required) in the past 3 months prior to screening.
4. Females of childbearing potential must have a negative urine or serum pregnancy test at screening and agree to continue use of an acceptable form of birth control throughout the duration of the study. Acceptable forms of birth control include oral, implant, injectable, and transdermal contraceptives; an intrauterine device; or other forms considered acceptable by the investigator. A female subject is eligible to participate if she is not pregnant, is not a woman or childbearing potential (WOCBP), or is a WOCBP who agrees to follow the contraceptive guidance above.
5. Post-pubertal males who agree to use an acceptable method of contraception for the duration of the study.
6. Subjects 18 years of age and older must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Subjects under the age of 18 years must be capable of giving assent (if age-appropriate), and/or they must have a guardian capable of providing consent.
7. Willing to comply with the protocol requirements.

Note: Reference to Appendix 3 can be located in the protocol

Exclusion Criteria:

1. Concomitant treatment at the time of screening or at any time during the study of either study wound (control or AGLE-102 treated) with local or systemic therapy other than standard of care treatments described in this protocol (i.e. local or systemic antimicrobials to control infection, topical anesthetic and oral analgesics if required). Concomitant treatment of non-study wounds with local therapy during the study is acceptable. Systemic treatment of RDEB wounds (except as noted for standard of care) during the study is not acceptable. Subjects unwilling to abstain from prohibited concomitant treatment of study wounds (treated or control) and/or systemic treatment of RDEB wounds during the study period are excluded.
2. Either study wound located within 6 inches of wounds treated concurrently with any other local therapy.
3. Clinical evidence of systemic infection.
4. History of bone marrow transplantation.
5. Diagnosed clinically significant autoimmune disease
6. Wound that extends across the fingers, toes, pubic or perineum region are excluded from being index wounds.
7. The subject has clinical evidence of an active infection at the wound site.
8. Current malignancy (including skin cancer), a life expectancy of < 2 years, or severe cardiopulmonary disease that restricts ambulation to the clinical facility.
9. History of coagulopathy.
10. Chronic use of systemic steroids or immunosuppressive agents.
11. Allergy to human albumin, streptomycin, or penicillin.
12. The subject is likely to be a recipient of tissue or organ transplantation.
13. Current history of alcohol or substance abuse or has a history of alcohol or substance abuse that required treatment within the previous 12 months.
14. History of poor compliance or unreliability.
15. Females who are pregnant, nursing, or planning a pregnancy during their participation in the study.
16. Concurrent participation in another investigational drug, biologic or device study that could confound study data.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events | 22 weeks
  Incidence of adverse events after single and repeat administrations of EVs
Wound healing improvement | 10 weeks
  Change in wound surface area relative to baseline compared with standard of care control

SECONDARY OUTCOMES:
Complete wound closure efficacy | 10 weeks
  Incidence of complete wound closure versus standard of care alone within 10 weeks
Time from baseline to complete wound closure | 22 weeks
  Time to wound closure versus standard of care alone
Scar quality improvement | 22 weeks
  Change from baseline in Patient and Observer Scar Assessment Scales. The min value is 1 and the max value is 10. The min value is normal skin and the max value is worst scar imaginable.
Pain relief efficacy | 22 weeks
  Change from baseline in patient reported pain using the Wong-Baker Faces Pain rating scale. The minimum value is value is 0 (no pain) and the maximum value is 10 (hurts worst).
Quality of Life Improvement | 22 weeks
  Change from baseline in patient reported Quality of Life scale. The minimum value is 0 (would does not affect you at all) and the maximum value is 5 (wound has maximum impact) on care, daily function, appearance, and concerns regarding others' reactions to the wound.

CONTACTS AND LOCATIONS:
Overall Officials: David T Woodley, MD, Principal Investigator — University of Southern California Dept of Dermatology
Locations (3):
- United States (3):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - USC /Norris Comprehensive Cancer Center University of Southern California, Los Angeles, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania